CLINICAL TRIAL: NCT03150095
Title: Health Coaching to Improve Self-Management in Thoracic Transplant Candidates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Cassie C. Kennedy, M.D., Associate Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-003921; K23HL128859 (NIH)
Record Dates: First submitted 2017-05-10; First posted 2017-05-11 (Actual); Results first posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-11

CONDITIONS: Self-management; Lung Transplant; Heart Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health coaching (Experimental): Patients will work with a health coach to improve self-management skills
  Interventions: Behavioral: Health coaching
- Control (No Intervention): Patients will receive usual pre-transplant education to improve self-management skills

INTERVENTIONS:
Behavioral: Health coaching — Patients will work with a health coach by telephone
  Arms: Health coaching

SUMMARY:
Ability to adhere to complex medical regimens is critical to achieving successful transplant outcomes, as non-adherent patients suffer graft failure and death following transplantation. Since potential recipients greatly exceed organ availability, identification of candidates who will adhere to complex post-transplant regimens is critically important and emphasized by practice guidelines. When selecting candidates for transplant, physicians try to subjectively predict post-transplant adherence because, although tools exist to measure current adherence, tools that reliably predict future adherence are lacking. Despite rigorous medical and psychosocial screening pretransplant, non-adherence rates are high following transplant. Therefore, the current approach for predicting future non-adherence is suboptimal, subjective, and greatly needs strategies for improvement.

Pre-transplant self-management abilities represent a marker of future adherence post-transplant. Assessing self-management as a means for predicting future adherence has been largely overlooked. Self-management is defined as "taking responsibility for one's own behavior and well-being" and consists of three management tasks: medical condition, emotions, and social roles. Self-management ability can be measured. However, self-management has not been systematically studied in heart and lung transplant patients. Fostering self-management abilities may improve post-transplant outcomes by optimizing not only adherence, but also proven pretransplant risk factors (e.g. frailty and obesity).Self-management abilities may be improved via behavioral interventions such as health coaching.Self-management represents a measurable criterion that could be utilized in pre-transplant screening and serve as a point of intervention for optimizing adherence and pre-transplant risk factors.The overall objective of the proposed research is to improve the knowledge gap regarding self-management (and thereby adherence) in transplant by qualitatively and quantitatively studying patient factors associated with self-management and testing an intervention that may improve self-management.

The investigators hypothesize: Individualized health coaching including strategies to address poor resilience, coping with uncertainty, frailty, and/or negative affect will be an effective therapeutic strategy at improving self-management while in the pre-transplant state.

Specific Aim: To test whether transplant candidates who receive pre transplant health coaching have greater improvement in self-management abilities.

The investigators will conduct a randomized, controlled pilot trial testing the effectiveness of health coaching versus usual care in a heart and lung transplant cohort on self-management abilities (SMAS-30).

DETAILED DESCRIPTION:
PROPOSED RESEARCH: Patients will be identified from the Mayo Clinic MN, heart and lung transplant waiting lists and approached for recruitment in the Transplant Clinic at one of their routine clinical (every 1 to 3 month) follow-up appointments or by phone or mail. Inclusion criteria: Aged 18 or older, consenting to research, and listed (active and temporarily inactive) or deferred for lung or heart transplantation at Mayo Clinic in Rochester, MN. Exclusion criteria: Patients will be excluded if ineligible for transplant, non-English speaking, non-verbal or extremely hard of hearing.

RESEARCH STRATEGY: This is a single-center, prospective, randomized, controlled, pilot study comparing the effect of a phone-based, health coaching intervention versus usual care on self-management. Methods: Initial encounter: Consented patients will be randomized using a random number generator. Intervention patients will be introduced to the intervention, and schedule the first phone meeting. Both intervention and control patients will undergo baseline assessments (see "data" below). Subsequent Coaching Intervention patients will be assigned a coach trained in motivational interviewing who will call the patient weekly for 12 weeks for a 15-30 minute intervention (based on the primary mentor's previous research). Briefly a health coaching protocol will be utilized to guide training and the delivery of intervention using open-ended questions, affirmations, reflections, and summaries (O.A.R.S.) and Elicit-Provide-Elicit (E-P-E) techniques. Coaching sessions will be recorded and externally monitored by an independent expert to assure treatment fidelity. A coaching intervention protocol will include collaborative goal setting and confidence rating regarding the patient's desired behavior change (and assessed risks). The control group will receive usual care. Both intervention and control patients will complete follow-up questionnaires and physiologic assessments at 12-16 weeks. Data: Baseline demographic, comorbidities, and transplant details will be abstracted. Daily physical activity measure by a gold standard activity monitor (Sensewear Armband, Body media, Pittsburgh,PA) will quantify daily steps, as well as total and active energy expenditure. Grip Strength: will be measured using a Jamar Digital Hand Held Dynamometer. Three serial measurements will be taken (using the dominant hand), averaged, and adjusted by gender and BMI using normative table. Gait Speed: self-selected walking speed will be timed over a distance of 15 ft (average of 3 adjusted for gender and height). Body composition scan: will determine fat-free mass (body composition). Height and weight will be recorded. Questionnaires: RISC-10, PANAS, MUIS, KCCQ, CRQ, FDI, CES-D, PHQ-2, GAD-2, SMAS-30, and SMAQ will be collected to assess hypothesized predictors of self-management. The primary outcome of the study is the effect of health coaching on self-management abilities SMAS-30 (sentinel of post- transplant adherence).

ANALYSIS PLAN: Sample size: This is a pilot and feasibility study. However, to inform our enrollment we have made the following calculations. Change in SMAS-30. A sample size of 25 in each group will have 80% power to detect an effect size of 0.81 using a two-group t-test with a 0.05 two-sided significance level, where effect size is the end of study difference in means between the two groups relative to the SD of the end of study measures, after adjusting for baseline and other factors. From the literature, we estimate an unadjusted end of study SD for SMAS-30 of 8.5.50 Whereas we do expect our intervention to impact SMAS-30, it is our clinical impression that without intervention, patients tend to exhibit similar patterns over time. Therefore, we expect the between-person variability in SMAS-30 to be at least as large as the variability in assessing SMAS-30 for the same person at different time points. If these two sources of variability were the same then they would both have a SD of 6.0, in particular the end of study SD for SMAS-30 would be 6.0 or less. With this SD, we would have power to detect a difference of 0.81x6.0=4.9. Thus, this pilot study is reasonably powered. Allowing for a 20% withdrawal rate (primarily due to transplantation during intervention), we will aim for a sample size of 30 per arm. Analysis plan: Demographic characteristics will be summarized by mean, median, SD and range (continuous variables) and counts and percents (categorical variables). Our primary variable will be end of study SMAS-30 (adjusting for baseline), which we will analyze using analysis of covariance (ANCOVA), estimating between group differences. Subgroup analysis will be performed by sex, ethnicity, and race as feasible. A similar procedure to that described above will be employed to impute data if necessary. Missing data and end of study SDs for SMAS-30, adjusting for baseline, will guide analysis and power calculations for future R01 studies. Secondary Outcomes will examine between group differences of changes in gait speed, activity levels, body composition, weights, and RISC-10, PANAS, MUIS, FDI, SMAQ, and KCCQ or CRQ measures to inform future R01 planning. A two-tailed p< 0.05 will be considered statistically significant. Post intervention focus groups/interviews of 5-7 participants will be conducted by the candidate to obtain patient feedback to refine the intervention for future R01.

ELIGIBILITY:
Inclusion Criteria:

* Subject is on heart or lung transplant waiting list

Exclusion Criteria:

* Under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cassie C Kennedy, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Health Coaching | Control
Started | 30 | 30
Completed | 21 | 28
Not Completed | 9 | 2
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 4 | 0
Not completed — unable or unwilling to continue health coaching | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Health Coaching | Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (8.1) | 55.0 (10.5) | 55.97 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 18 | 18 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 25 | 24 | 49
  Unknown or Not Reported | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 29 | 26 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Score on Baseline Self-Management Ability Scale (SMAS-30) [Mean (Standard Deviation); unit: score on a scale] — The 30 Item Self-Management Ability Scale (SMAS-30) measures self-management based on questions from 6 subsets of Taking Initiatives, Investment Behavior, Variety, Multifunctionality, Self-efficacy, and Positive Frame of Mind. These are totaled into a scale ranging from 0-100. Higher scores indicate better self-management ability.
  score on a scale | 70.31 (13.49) | 70.74 (11.68) | 70.53 (12.51)

OUTCOME MEASURES:

1. Primary Outcome: Score on Follow-up Self-Management Ability Scale (SMAS-30)
Description: The 30 Item Self-Management Ability Scale (SMAS-30) measures self-management based on questions from 6 subsets of Taking Initiatives, Investment Behavior, Variety, Multifunctionality, Self-efficacy, and Positive Frame of Mind. These are totaled into a scale ranging from 0-100. Higher scores indicate better self-management ability.
Time Frame: 12-16-week follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Coaching | Control
Number analyzed (Participants) | 21 | 28
score on a scale | 75.06 (17.01) | 71.47 (11.09)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Health Coaching | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 1/30
Serious Adverse Events (participants affected / at risk) | 1/30 | 1/30
Other Adverse Events (participants affected / at risk) | 1/30 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Health Coaching (N=30) | Control (N=30)
Unplanned Hospital Admission (Surgical and medical procedures) | 1 (1) | 0 (0) — Not related to study
Fatal Automobile Accident (Social circumstances) | 0 (0) | 1 (1) — by motor vehicle accident
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Health Coaching (N=30) | Control (N=30)
Respiratory symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/95/NCT03150095/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT03150095/SAP_001.pdf
  • Informed Consent Form (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/95/NCT03150095/ICF_002.pdf